CLINICAL TRIAL: NCT02181998
Title: A Phase IIIb-IV, Randomised, Open Label Trial on Efficacy and Safety of 2 Parallel Groups: Full Dose Tenecteplase Combined With Unfractionated Heparin or Enoxaparin in Acute Myocardial Infarction in the Prehospital Setting (ASSENT 3 Plus) ASSENT 3 Plus Was a Satellite Study to ASSENT 3 (Main Study) ASSENT (ASsessment of the Safety and Efficacy of New Thrombolytic Regimens)
Brief Title: A Trial on Efficacy and Safety of Full Dose Tenecteplase Combined With Unfractionated Heparin (UFH) or Enoxaparin in Acute Myocardial Infarction (AMI) in the Prehospital Setting
Acronym: ASSENT 3 Plus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1123.11
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Enoxaparin

ARMS (2):
- tenecteplase + unfractioned heparin (Active Comparator)
  Interventions: Drug: Full dose tenecteplase; Drug: Unfractioned heparin
- tenecteplase + enoxaparin (Experimental)
  Interventions: Drug: Full dose tenecteplase; Drug: Enoxaparin

INTERVENTIONS:
Drug: Full dose tenecteplase
Drug: Unfractioned heparin
  Arms: tenecteplase + unfractioned heparin
Drug: Enoxaparin
  Arms: tenecteplase + enoxaparin

SUMMARY:
The primary objective of ASSENT 3 Plus (the same as for ASSENT 3) was to evaluate the safety and efficacy of full dose tenecteplase combined with unfractionated heparin (UFH, group A) and full dose tenecteplase combined with enoxaparin (ENOX, group B). An additional objective in ASSENT 3 Plus was to describe the different time intervals in the prehospital phase.

ELIGIBILITY:
Inclusion Criteria:

* Onset of symptoms of AMI within six hours prior to randomisation
* A 12-lead ECG with one of the following: ST-segment elevation ≥ 0.1 millivolt (mV) in two or more limb leads, or ≥ 0.2 mV in two or more contiguous precordial leads indicative of AMI, or left bundle-branch block
* Age ≥ 18
* Informed consent received

Exclusion Criteria:

* Hypertension defined as blood pressure (BP) > 180/110 mmHg (systolic blood pressure (SBP) 180 mmHg and/or diastolic blood pressure (DBP) > 110 mmHg) on repeated measurements during current admission prior to randomisation
* Use of abciximab (ReoPro ®) or other glycoprotein-IIb/IIIa antagonists within the preceding seven days
* Major surgery, biopsy of a parenchymal organ, or significant trauma within two months
* Any minor head trauma and any other trauma occurring after onset of the current myocardial infarction (MI)
* Any known history of stroke or transient ischaemic attack or dementia
* Any known structural damage of the central nervous system
* Prolonged cardiopulmonary resuscitation (> 10 min) in the previous two weeks
* Current oral anticoagulation
* Standard UFH (heparin sodium) > 5000 international units (IU), or a subcutaneous (SC) therapeutic dose of any low molecular weight heparin (LMWH) within six hours of randomisation
* Known thrombocytopenia (prior platelet count below 100 000 cells/μL (100 x 10**9/L))
* Known renal insufficiency (prior S-creatinine > 2.5 mg % (> 220 μmol/L) for men and 2.0 mg % (> 175 μmol/L)) for women
* Pregnancy or lactation, parturition within the previous 30 days. Women of childbearing potential had to have a negative pregnancy test, or use a medically accepted method of birth control
* Treatment with an investigational drug under another study protocol in the past seven days
* Previous enrolment in this study
* Known sensitivity to tenecteplase, tissue plasminogen activator (tPA), abciximab, heparin or LMWH
* Any other condition that the investigator felt would place the patient at increased risk if the investigational therapy was initiated (e.g. known haemorrhagic diathesis, acute pericarditis and/or subacute bacterial endocarditis, acute pancreatitis, severe hepatic dysfunction, diabetic haemorrhagic retinopathy or other haemorrhagic ophthalmic conditions, active peptic ulceration, arterial aneurysm and known arterial/venous malformation, neoplasm with increased bleeding risk)
* Inability to follow protocol and comply with follow-up requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1606 (Actual)
Dates: Start 2000-07; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Composite endpoint: 30-day mortality or in-hospital reinfarction or in-hospital refractory ischemia or in-hospital intracranial hemorrhage (ICH) or in-hospital major bleedings (other than ICH) | Up to 30 days after discharge from hospital
Composite endpoints: 30-day mortality or in-hospital reinfarction or in-hospital refractory ischemia | Up to 30 days after discharge from hospital